CLINICAL TRIAL: NCT05305313
Title: Evaluation of Propofol Dosing Based on Total Body Weight Versus Adjusted Body Weight in Obese Patients Receiving Total Intravenous Anaesthesia With Automated Closed-Loop Anaesthesia Delivery System: A Randomized Controlled Study
Brief Title: Evaluation of Propofol Dosing Based on Total Body Weight Using Closes-loop Anaesthesia Delivery System
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Nitin Sethi, DNB, Principal Investigator, Sir Ganga Ram Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: EC/01/22/1992
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Obesity, Morbid; Anesthesia; Propofol
MeSH Terms: conditions — Obesity, Morbid | interventions — Propofol

STUDY DESIGN:
Intervention Model Description: Forty six- patients of either sex, and schedule for laparoscopic and non-laparoscopic surgery of more than 60-minutes duration will be randomly divided into two groups of 23 each patients:
  Group-I [TBW group, n=23]: Patients in this group will receive maintenance propofol calculated using total body weight (TBW).
  Group-II [ABW group, n=23]: Patients in this group will receive maintenance propofol calculated using adjusted body weight (ABW).
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will be blinded to the type of anaesthesia intervention. The attending anaesthesiologist will however not be blinded to the technique utilized to administer GA and recovery immediately after extubation inside the OR. The postoperative patient recovery profile will be evaluated by an independent assessor blinded to the technique of GA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total Body Weight group (Active Comparator): Anesthesia will be induced and maintained with Propofol administered by CLADS which will be set to deliver Propofol according to total body weight (TBW). A BIS-value of 50 will be used as the target for induction and maintaenance of anesthesia.
  Interventions: Drug: Propofol
- Adjusted Body Weight group (Active Comparator): Anesthesia will be induced and maintained with Propofol administered by CLADS which will be set to deliver Propofol according to adjusted body weight (ABW). A BIS-value of 50 will be used as the target for induction and maintenance of anesthesia.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol delivery will be controlled using automated closed loop anaesthesia delivery system which will control propofol delivery rate to consistent anaesthetic depth (BIS-50) feedback from the patient.
  Arms: Total Body Weight group
Drug: Propofol — Propofol delivery will be controlled using automated closed loop anaesthesia delivery system which will control propofol delivery rate to consistent anaesthetic depth (BIS-50) feedback from the patient.
  Arms: Adjusted Body Weight group

SUMMARY:
The pharmacokinetic profile of various drugs is altered in obese patients especially those administered by the intravenous route. Propofol is the commonly used intravenous anesthetic agent for induction and maintenance of anaesthesia as part of total intravenous anaesthesia (TIVA) regimen. A major concern with propofol dosing based on total body weight (TBW) in obese patients is disproportionate drug administration leading to undue drug accumulation in body with a potential to overdosing, delayed recovery from anaesthesia, and adverse hemodynamic outcome. Studies on propofol dosing based on various weight scalars have recommended that lean body weight (LBW) should be used for calculating bolus dose during anaesthesia induction and TBW or adjusted body weight (ABW) for arriving at an infusion dose required for maintenance of anesthesia. Although propofol delivery based on dose calculated by TBW has been well researched the evidence for propofol delivery based on dose calculated by ABW is lacking.

Recent advance in the delivery of propofol has been the development of computer controlled anaesthesia delivery systems. These devices deliver propofol based on patient's frontal cortex electrical activity as determined by bispectral index (BIS). Evaluation of anaesthesia delivery by these systems has shown that they deliver propofol and maintain depth of anaesthesia with far more precision as compared to manual administration. One such indigenously developed computer controlled anaesthesia delivery system is the closed loop anesthesia delivery system (CLADS). CLADS functions on control of processed EEG response parameter captured from anesthetized patients with the help of a BIS- monitor, which is continuously fed into an automated drug infusion pump. The infusion pump then accordingly delivers the anesthetic drug to the patients based on pharmacodynamic requirements. The investigators plan to evaluate the propofol maintenance dose requirement based on TBW versus ABW using CLADS for propofol delivery.

DETAILED DESCRIPTION:
Propofol is the most used intravenous agent for induction and maintenance of anaesthesia as part of total intravenous anaesthesia (TIVA) regimen.

In the morbidly obese, various factors, such as, increased body fat content, lean body weight, cardiac output, total blood volume, and alterations in regional blood flow; which adversely/unpredictably affect the volume of distribution, clearance and elimination of intravenous anesthetic drugs, thereby making administration of TIVA difficult to control.

A major concern with propofol dosing based on total body weight (TBW) in the obese patients is disproportionate drug administration leading to undue drug accumulation in body with potential overdosing, delayed recovery from anaesthesia, and adverse hemodynamic outcome. Studies on propofol dose regimen for TIVA recommended that LBW should be used for calculating bolus dose during induction of anaesthesia and TBW or ABW for arriving at a infusion dose required for maintenance of anaesthesia.

Propofol requirement for induction of anaesthesia is based on LBW is especially relevant for the morbidly obese patients as because their surplus fat mass increases volume of distribution of propofol, which, in the face of decreased blood flow to adipose tissue; imposes the burden of potential drug accumulation. This may result in increased drug delivery to non-adipose tissue during induction of anaesthesia and possibly leading to undesirable rarefaction of depth-of-anaesthesia and attendant adverse haemodynamic effects.

Conversely, during the maintenance phase of propofol TIVA, the volume of distribution and clearance of propofol increases and correlates linearly with TBW. In this respect, controlling propofol delivery in the morbidly obese with Eleveld allometric PK model, which utilizes TBW as weight parameter; has been found to be superior to other models that employs other weight dosing scalars.

The use of ABW in Schnider and Marsh model takes into consideration drug distribution to lean tissues as well as a proportion to the body fat weight, thus accounting for lipid solubility dynamics of propofol. ABW is calculated by adding 40% excess fat weight (FW) to IBW.

In obese patients propofol delivery using the Eleveld allometric PK model by incorporating TBW has been found to be superior to other models using other dosing scalars.

Target-controlled infusion (TCI) forms the core of standard-of-care method used for administration of propofol TIVA. TCI system typically includes a microprocessor-controlled syringe pump that is designed to achieve a defined plasma concentration of the drug based on patient response and multi-compartment pharmacokinetic (PK) model.

While TCI systems are designed to deliver propofol at a rate based on a predetermined plasma concentration, they do not take into consideration patient's pharmacodynamic profile. Hence, it is difficult to determine whether the target plasma concentration achieved has produced adequate anaesthesia depth. In the absence of reliable depth of anaesthesia monitors, during the maintenance phase of propofol TIVA, the desired plasma concentration achieved may either result in intraoperative awareness due to under-dosing or delayed recovery from anaesthesia because of over-dosing.

Currently, an array of research on automated propofol delivery using computer-controlled closed loop anaesthesia delivery systems which deliver propofol based on patient's frontal cortex electrical activity as determined by bispectral index (BIS); have amply exhibited that these systems deliver propofol and maintain depth of anaesthesia with far more precision as compared to manual administration.

Liu et al used a BIS-guided dual loop anaesthesia delivery system to determine requirement of propofol and remifenatnil in the obese versus lean patients. The propofol delivery was controlled by a closed loop set through TCI pump. Propofol was delivered with dose calculation by TBW and based on the Schnider model. The propofol dosage delivered as per TBW in real-time was analyzed post hoc on a IBW scale. The propofol requirements for induction and maintenance based on TBW was equivalent both in obese and lean patients.

CLADS is a BIS-guided automated closed-loop anaesthesia delivery system developed by Puri, which delivers propofol using a non-TCI infusion pump. This system uses a control algorithm that is based on the relationship between diverse rates of propofol infusion and BIS variable. CLADS regulates the propofol infusion rate to maintain a predetermined BIS target (BIS=50) and is independent of plasma propofol concentration status. CLADS is uniquely versatile in that it can calculate propofol dosage delivered both on basis of TBW or IBW.

Whereas, in a study comparing CLADS administered propofol versus desflurane-GA in morbid obese patients undergoing bariatric surgery (unpublished data) the propofol maintenance dosage based on ABW was 5.5 + 1.3 mg kg-1 h-1; Liu et al reported a median propofol consumption of 5.2 [4.1, 6] mg kg-1 h-1 with their dual-loop closed loop anaesthesia delivery system that also utilized TBW based administration of propofol and remifentanil. In both the study, BIS was used as an input control actuator to close the feedback loop joining the patient, the delivery system, and the infusion flow system.

Although maintenance of propofol TIVA based on TBW is well established, the dosing schedule based on ABW is not well explored. Since the ABW takes into consideration a certain percentage of FW in addition to IBW and not the complete FW as in TBW, we hypothesize that propofol dosing using ABW will result in lower propofol requirement as compared to TBW for maintaining equivalent anesthetic depth. Since CLADS gives an objective assessment of propofol dose delivered and anaesthesia depth consistency, this randomized study aim to compare the maintenance requirements of propofol in obese patients given propofol dosing based on TBW versus ABW

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status II/III
2. laparoscopic and non-laparoscopic surgery of more than 60-minutes duration
3. Body mass index > 35kg/m2

Exclusion Criteria:

1. Cardiovascular disorders (uncontrolled hypertension, Atrio-ventricular block, sinus bradycardia, congenital heart disease, reduced LV compliance & diastolic dysfunction)
2. Neurological disorders (previous neurosurgery, psychiatric disorders, autonomic nervous system disorders- orthostatic hypotension, transient ischemic attacks)
3. Hepato-renal insufficiency
4. Uncontrolled diabetes mellitus
5. Known allergy/hypersensitivity to study drug
6. Pulmonary dysfunction (restrictive /obstructive lung disease)
7. Acute/chronic drug dependence/substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2026-11-04 (Estimated); Study Completion 2026-11-10 (Estimated)

PRIMARY OUTCOMES:
Propofol Maintenance Dose (mg/kg/hour) | From start of anesthesia till 5- minutes post skin closure
  Propofol required for maintenance of anaesthesia based on total body weight versus adjusted body weight

SECONDARY OUTCOMES:
Anaesthesia Depth consistency | From start of anesthesia till 5- minutes post skin closure
  Percentage of the total valid CLADS time during which the BIS remained + 10% of the target BIS value of 50.
Performance characteristic of propofol delivery system | From start of anesthesia till 5- minutes post skin closure
  It will be determined using the Varvel criteria parameter :median performance error (MDPE). This parameter is calculated by the computer software which analyses the intraoperative BIS data. This parameter have no unit of measurement. Its just a abstract number
Performance characteristic of propofol delivery system | From start of anesthesia till 5- minutes post skin closure
  It will be determined using the Varvel criteria parameter: median absolute performance error (MDAPE).This parameter is calculated by the computer software which analyses the intraoperative BIS data. This parameter have no unit of measurement. Its just a abstract number.
Performance characteristic of propofol delivery system | From start of anesthesia till 5- minutes post skin closure
  It will be determined using the Varvel criteria parameter: wobble. This parameter is calculated by the computer software which analyses the intraoperative BIS data. This parameter have no unit of measurement. Its just a abstract number.
Performance characteristic of propofol delivery system | From start of anesthesia till 5- minutes post skin closure
  It will be determined using the Varvel criteria parameter: global score. It is calculated using the formula Median absolute performance error + wobble / percentage of the anesthesia time during which the BIS remained +/- 10 of the target BIS of 50. This parameter have no unit of measurement. Its just a abstract number.
Intra-operative heart Rate (beats per minute) | From beginning of anaesthesia till 10 hours intraoperatively
  Comparison of intra-operative heart rate between the study arms will be done
Intra-operative systolic , diastolic, and mean blood pressure (mmHg) | From beginning of anaesthesia till 10 hours intraoperatively
  Comparison of intra-operative blood pressure- systolic, diastolic, and mean blood pressure between the study arms will be done
Early recovery from anaesthesia | From beginning of anaesthesia till 30-minutes postoperatively
  Time taken by the patient to open his/her eyes after discontinuation of anaesthesia will be noted
Early recovery from anaesthesia | From beginning of anaesthesia till 30-minutes postoperatively
  Time taken for tracheal extubation after discontinuation of anaesthesia will be noted
Postoperative sedation | From end of anaesthesia till 24-hours postoperatively
  Will be assessed using Modified Observer's assessment of alertness/sedation scale. The scale has a maximum value of '5', which refers to a fully awake patient and a minimum value of '0' which refers to a deeply sedated patient.
Intraoperative awareness | From the end of anaesthesia till 48-hours, postoperatively
  Will be assessed using modified brice questionnaire. The questionnaire has a set of '5' questions, if answer to any of the question is in affirmative then it is suggestive of intraoperative awareness

CONTACTS AND LOCATIONS:
Overall Officials: Goverdhan D Puri, MD, PhD, Study Director — Post Graduate Institute of Medical Education & Research, Chandigarh, India; Jayashree Sood, MD, FFRCA, PGDHHM, FICA, Study Chair — Sir Ganga Ram Hospital, New Delhi, INDIA
Locations (1):
- Nitin Sethi, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No